CLINICAL TRIAL: NCT06259851
Title: rTMS-enhanced Psychotherapy for Borderline Personality Disorder
Acronym: rTMS-DBT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masarykova Univerzita (Other)
Collaborators: Brno University Hospital (Other); Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NU23-04-00472
Record Dates: First submitted 2023-10-09; First posted 2024-02-14 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Borderline Personality Disorder
Keywords: Dialectical behavioral therapy; Repetitive transcranial magnetic stimulation; Borderline personality disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: Allocation to the Active rTMS/Sham rTMS group is randomized.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- rTMS-DBT group (Experimental): Patients receiving combined DBT and active prefrontal rTMS treatment
  Interventions: Behavioral: Dialectical behavioral therapy program; Device: Prefrontal rTMS treatment
- Sham-DBT group (Active Comparator): Patients receiving combined DBT and sham rTMS treatment
  Interventions: Behavioral: Dialectical behavioral therapy program; Device: Sham rTMS sessions
- rTMS-only group (Active Comparator): Patients receiving only active prefrontal rTMS treatment
  Interventions: Device: Prefrontal rTMS treatment
- sham-only group (Sham Comparator): Patients receiving only sham rTMS treatment
  Interventions: Device: Sham rTMS sessions

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy program — Dialectical behavioral therapy (DBT) program with all the standard DBT modules (individual therapy 1 hour per week, skills group 3 hours per week, phone coaching, and therapist consultation team 1,5 hour per week). The program takes 24 weeks in total comprising two 12-week runs of skills training. The program will be precluded with 4 individual sessions of pretreatment before the start of the main program part.
  Arms: Sham-DBT group; rTMS-DBT group
Device: Prefrontal rTMS treatment — rTMS will be performed by DuoMag XT with 70BF cool coil. Patients will undergo 15 daily stimulation sessions during a period of three weeks with one session each working day. Each session consists of 20 trains with 100 pulses (10 seconds for train). Inter-train interval will be 30 seconds. Gradual titration of the individual resting motor threshold (RMT) will apply, meaning probands will undergo first session with 90% RMT intensity, second session with 100% RMT intensity, third session with 110% RMT intensity. All the following sessions will use the final 120% RMT intensity. In case a session is left out because of any reason, the total duration of treatment will be prolonged by one day, so that the total number of sessions underwent is the same in all patients. Patients will receive 2000 pulses during one session (total 30000 pulses during the whole procedure) with 10 Hz frequency.
  Arms: rTMS-DBT group; rTMS-only group
Device: Sham rTMS sessions — Sham TMS will be performed by sham coil that looks identical to DuoMag XT in the active group. Patients will undergo 15 daily sham stimulation sessions during a period of three weeks with one session each working day. Each session consists of 20 trains with 100 pulses (10 seconds for train). Inter-train interval will be 30 seconds.
  Arms: Sham-DBT group; sham-only group

SUMMARY:
This project assesses the effectiveness and lasting impact of combining Dialectical Behavioral Therapy (DBT) with prefrontal repetitive transcranial magnetic stimulation (rTMS) in patients with borderline personality disorder.

DETAILED DESCRIPTION:
The proposed project aims to evaluate the effectiveness of combining Dialectical Behavioral Therapy (DBT) with prefrontal repetitive transcranial magnetic stimulation (rTMS) in individuals with borderline personality disorder (BPD). The study includes four groups of patients: 1) DBT combined with active prefrontal rTMS treatment (rTMS-DBT group), 2) DBT combined with sham rTMS treatment (sham-DBT group), 3) active prefrontal rTMS treatment only (rTMS-only group), and 4) sham rTMS treatment only (sham-only group). The study will include assessments conducted before (T1) and after the rTMS treatment (T2) composed of self-reported questionnaires, clinical interviews assessing self-harming behavior and healthcare utilization, ecological momentary assessment of emotional variability, functional magnetic resonance imaging (fMRI) during emotional task, and control clinical EEG measurements. Follow-up measurements will be conducted at T3 (three months after rTMS), and for DBT group also at T4 (six months after rTMS), and T5 (twelve months after rTMS) for to track long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of borderline personality disorder according to Diagnostic and Statistical Manual 5th Edition (DSM-5) criteria (rated by Structured Clinical Interview for DSM-5 for Personality Disorders, BPD section)
* minimum age 16, informed consent of the patient
* informed consent of patient's legal representative in case of patients under age 18

Exclusion Criteria:

* neurological disorder
* comorbid affective disorder or schizophrenia-related disorder
* intelligence quotient<70
* contraindications for MRI measurement
* contraindication for rTMS treatment
* pregnancy

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — cisgender female
Enrollment: 60 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Decrease of borderline symptoms | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  significant decrease of symptoms measured by Borderline Symptoms List-23
Decrease of impulsivity | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  significant decrease of impulsivity measured by UPPS-P questionnaire
Increase of emotion regulation | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  significant increase of emotion regulation measured by Difficulties in emotion regulation scale (minimum: 22, maximum: 87, higher score means better outcome)
Decrease of self-reported depression symptoms | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  significant decrease of depression symptoms measured by Beck Depression Inventory II
Decrease of depression symptoms clinical ranking | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  significant decrease of depression symptoms measured by Montgomery-Asberg Depression Rating Scale clinical rating
Decrease of anxiety | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  significant decrease of anxiety symptoms measured by Beck Anxiety Inventory
Decrease of dissociation symptoms | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  significant decrease of dissociation symptoms measured by Multiscale dissociation inventory
Increased regulation of amygdala during fMRI neurofeedback | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3) in all groups and additionally 24 weeks after baseline (T4) in DBT group
  fMRI neurofeedback will be used to measure the participants' ability to influence their amygdala activity. fMRI neurofeedback is a method which enables measuring, computing, and displaying the current blood oxygen level-dependent (BOLD) signal level in a selected brain area. The ability of the participants to voluntarily regulate the target area activity using the feedback presentation is measured. Specifically, pictures arousing negative emotions will be presented to participants in the MR scanner together with a scale showing the current level of their right amygdala activity and participants will be instructed to decrease the scale as much as possible by regulating down their emotion (regulation condition). As a controlled condition to regulation condition, passive viewing of the negative pictures will be included (view condition).
Decreased brain emotional reactivity | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3) in all groups and additionally 24 weeks after baseline (T4) in DBT group
  Hariri task (fMRI emotional processing task) in fMRI will be used to measure brain correlates of emotional reactivity. The task includes 2 experimental categories: 1. emotional faces and 2. emotional social scenes which reliably evoke emotional responses, and 1 control baseline condition of geometric shapes. Further, each experimental category will include three condition: negative pictures, positive pictures, and neutral pictures. Contrast of emotional conditions against neutral conditions of the same type and against control condition will be used to track the neural correlates of emotional reactivity and processing.
Decreased impulsivity in Go/No-Go task in fMRI | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3) in all groups and additionally 24 weeks after baseline (T4) in DBT group
  fMRI Go/No-Go task will be displaying 2 experimental conditions (presenting letter A or X), where participant is asked to react with a button only in first condition (Go condition), while remain passive during the second condition (NoGo condition). The task is designed to measure impulsivity and brain correlates during inhibition.
Decrease of emotional variability | Baseline (T1), after 3 weeks (T2), 12 weeks after baseline (T3), 24 weeks after baseline (T4) in all groups and additionally 48 weeks after baseline (T5) in DBT group
  Measured by ecological momentary assessment (EMA) implemented as an questionnaire accessible through participant's smartphone via application ExpiWell. Participants will receive notifications reminding to fill out the questionnaire every hour (in random times during the hour) between 9 am and 9 pm for two days. Participants will be asked about their current experienced emotion and its intensity. Additional questions on self-harm and suicidal thoughts intensity during the day and whether a self-harming incident has occurred during the day will be sent at 9 pm on both days.
Decrease in sef-harming behavior and medical care usage | Recorded for the past 6 months (at the beginning and after 48 weeks) or in the past three months (after 12 weeks and after 24 weeks)
  During an interview with a clinician, participants will be asked about the number of self-harming incidents and suicidal attempts and the number of crisis medical care usage and number of days spent in psychiatric hospitalization in the past 6 months or in the past three months.

CONTACTS AND LOCATIONS:
Overall Officials: Libor Ustohal, prof, Ph.D., Principal Investigator — University Hospital Brno
Locations (1):
- Department of Psychiatry, University Hospital Brno and Faculty of Medicine, Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All IPD in anonymized form that underlie results will be shared on request after approval of principal investigator.
Time Frame: 1 year after publication of the results.
Access Criteria: Access requests can be submitted by email to Central contact person: Pavla Linhartová.